CLINICAL TRIAL: NCT06026839
Title: Longitudinal Study on the Quality of Life of Pediatric Patients After Hematopoietic Stem Cell Transplantation and Its Influencing Factors
Brief Title: Longitudinal Study on the QoL of Pediatric Patients After HSCT and Its Influencing Factors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-339-01
Record Dates: First submitted 2023-06-21; First posted 2023-09-07 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Thalassemia Major; Acute Leukemia
Keywords: hematopoietic stem cell transplantation; children; quality of life
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Conventional nursing — Conventional nursing

SUMMARY:
Objective: To longitudinally track the dynamic changes in the survival quality of pediatric patients after hematopoietic stem cell transplantation at different time points within 1 year post-transplantation, analyze the influencing factors of survival quality at each time point, identify independent risk factors that can be intervened, provide reference for medical staff to recognize survival quality problems early, guide the dynamic management of clinical survival quality, and formulate continuation care management plans.

Methods: This study adopted a repeated measurement study design. A total of 250 pediatric patients who underwent hematopoietic stem cell transplantation in three tertiary hospitals in Guangdong Province from August 2023 to December 2025 and met the research standards were selected as the research subjects. The "Childhood Health Assessment Questionnaire Transplant Module 3.0 Chinese Version" was used to evaluate the survival quality of the patients at six time points: 1 week before pre-treatment (T0), the day of stem cell infusion (T1), 1 month (T2), 3 months (T3), 6 months (T4), and 1 year (T5) after transplantation. Statistical methods for repeated measures were used to analyze the relevant information, and mixed-effect linear models were used to analyze the influencing factors of survival quality at the six time points, and to identify independent risk factors.

DETAILED DESCRIPTION:
Objective: longitudinal tracking hematopoietic stem cell transplantation in 1 years after transplantation in different time points of the quality of life dynamic change trajectory, analyze the factors of quality of each time point, looking for independent risk factors for intervention, early identification of life quality for medical staff, guide the clinical quality of life dynamic management and continuation of nursing management plan to provide reference basis. Methods: In this study, 250 children with routine HSCT transplantation were selected from August 2023 to December 2025 (T1), 1 month (T2), 3 months after transplantation, 1 year after transplantation (T5). Statistical analysis of relevant information was performed using repeated measures, and the influencing factors of QOL at six time points were used to identify their independent risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. children aged between 0 and 18 years old who will receive a stem cell infusion
2. conscious, have a certain level of cognitive ability and be able to express their physical and psychological state accurately
3. If the child is under 8 years old, their caregiver should have a primary school or higher education level with sufficient reading comprehension and expression abilities
4. both the child and the legal guardian are informed and consent to participate in the study

Exclusion Criteria:

1. the child has a history of mental illness
2. the child has severe organ failure or other serious complications involving the heart, brain, lungs, liver, kidneys, and other organs

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a planned study on hematopoietic stem cell transplantation for children aged between 0 and 18 years old who will receive a stem cell infusion. The children must be conscious, have a certain level of cognitive ability and be able to express their physical and psychological state accurately. If the child is under 8 years old, their caregiver should have a primary school or higher education level with sufficient reading comprehension and expression abilities. It is important that both the child and the legal guardian are informed and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PedsQL™ 3.0 | 2023.6.30-2024.12.31
  the Chinese mandarin version of PedsQL™ 3.0 transplant module

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Since the study involves vulnerable populations, consent from guardians must be obtained before further data sharing can take place. This is to protect research subjects and adhere to ethical guidelines. During the process of data sharing, strict control over data usage is needed to ensure confidentiality and security of the data.

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT06026839/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT06026839/SAP_001.pdf